CLINICAL TRIAL: NCT02947685
Title: A Randomized, Open Label, Phase III Trial to Evaluate the Efficacy and Safety of Palbociclib + Anti-HER2 Therapy + Endocrine Therapy vs. Anti-HER2 Therapy + Endocrine Therapy After Induction Treatment for Hormone Receptor Positive (HR+)/HER2-Positive Metastatic Breast Cancer
Brief Title: Randomized, Open Label, Clinical Study of the Targeted Therapy, Palbociclib, to Treat Metastatic Breast Cancer
Acronym: PATINA
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Alliance Foundation Trials, LLC. (Other)
Collaborators: Pfizer (Industry); GBG Forschungs GmbH (Other); Fondazione Michelangelo (Other); PrECOG, LLC. (Other); Breast Cancer Trials, Australia and New Zealand (Other); Syneos Health (Other); SOLTI Breast Cancer Research Group (Other); UNICANCER (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: AFT-38
Record Dates: First submitted 2016-10-26; First posted 2016-10-28 (Estimated); Results first posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: HER-2 Positive Breast Cancer; Estrogen Receptor Positive Breast Cancer
Keywords: breast cancer; malignant tumor of the breast; HER2+; HR+; metastatic breast cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — palbociclib; Trastuzumab; pertuzumab; Letrozole; Anastrozole; exemestane; Fulvestrant

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (Experimental): Palbociclib 125 mg daily + AntiHER2 Therapy (trastuzumab/pertuzumab) q3wks + Endocrine Therapy (letrozole, anastrozole, exemstane OR fulvestratnt) until confirmed disease progression
  Interventions: Drug: palbociclib; Drug: trastuzumab; Drug: pertuzumab; Drug: letrozole; Drug: Anastrozole; Drug: Exemestane; Drug: Fulvestrant
- Arm B (Active Comparator): AntiHER2 Therapy (trastuzumab/pertuzumab) q3wks + Endocrine Therapy (letrozole, anastrozole, exemstane OR fulvestrant) until confirmed disease progression
  Interventions: Drug: pertuzumab; Drug: letrozole; Drug: Anastrozole; Drug: Exemestane; Drug: Fulvestrant

INTERVENTIONS:
Drug: palbociclib — o Starting dose: 125 mg capsule taken orally once per day for 21 days followed by 7 days off to complete 28 day cycle. Dose reductions: 100 mg, 75 mg. allowed. Number of Cycles: until progression or unacceptable toxicity develops
  Other Names: Ibrance
  Arms: Arm A
Drug: trastuzumab — Patients must have received a minimum of 4 and maximum of 8 cycles of induction therapy prior to randomization to Arm A or B, at which point they will continue on antiHER2 therapy and endocrine therapy, with or without palbociclib. Trastuzumab dosing will be determined based on a loading dose of 8mg trastuzumab/kg body weight for Q3WK dosing schedules or a maintenance dose of 6mg/kg trastuzumab/kg dosing weight for Q3WK dosing schedules. Loading dose will be administered on Cycle 1, Day 1.
  Other Names: Herceptin
  Arms: Arm A
Drug: pertuzumab — Patients must have received a minimum of 4 and maximum of 8 cycles of induction therapy prior to randomization to Arm A or B, at which point they will continue on antiHER2 therapy and endocrine therapy, with or without palbociclib.Pertuzumab will be administered at a loading dose of 840 mg infusion and then at a maintenance dose of 420 mg q3wks. If patient is within 5 weeks of receiving loading dose at Cycle 1, Day 1, patient may start with maintenance dose of 420 mg.
  Other Names: Perjeta
Drug: letrozole — There are several allowed endocrine treatment agents for Arm A and Arm B of this study. Administration is performed on an outpatient, self-administration basis according to local requirements and local standard practice. Endocrine treatment may have started before the patient enters the study. Agents will be administered at the discretion of principal investigator as well as according to standard institutional or regional practice. Recommended dosing regimen for letrozole oral therapy is 2.5 mg orally, once a day.
  Other Names: Femara
Drug: Anastrozole — There are several allowed endocrine treatment agents for Arm A and Arm B of this study. Administration is performed on an outpatient, self-administration basis according to local requirements and local standard practice. Endocrine treatment may have started before the patient enters the study. Agents will be administered at the discretion of principal investigator as well as according to standard institutional or regional practice. Recommended dosing regimen for anastrozole is 1 mg orally, once a day.
  Other Names: Arimidex
Drug: Exemestane — There are several allowed endocrine treatment agents for Arm A and Arm B of this study. Administration is performed on an outpatient, self-administration basis according to local requirements and local standard practice. Endocrine treatment may have started before the patient enters the study. Agents will be administered at the discretion of principal investigator as well as according to standard institutional or regional practice. Recommended dosing regimen for exemestane is 25 mg orally, once a day.
  Other Names: Aromasin
Drug: Fulvestrant — There are several allowed endocrine treatment agents for Arm A and Arm B of this study. Administration is performed on an outpatient, self-administration basis according to local requirements and local standard practice. Endocrine treatment may have started before the patient enters the study. Agents will be administered at the discretion of principal investigator as well as according to standard institutional or regional practice. Recommended dosing regimen for Fulvestrant is 250 mg injections on Day 1 and Day 15 of Cycle 1, and q4weeks thereafter.
  Other Names: Faslodex

SUMMARY:
The primary objective of this study is to demonstrate that the combination of palbociclib with anti-HER2 therapy plus endocrine therapy is superior to anti-HER2-based therapy plus endocrine therapy alone in improving the outcomes of subjects with hormone receptor-positive, HER2+ metastatic breast cancer.

DETAILED DESCRIPTION:
Subjects will be randomized into one of two treatment arms following minimum of 4 and maximum of 8 cycles of induction treatment with anti-HER2 therapy. Arm A subjects will receive the experimental therapy, palbociclib, in addition to their current anti-HER2 therapy and endocrine therapy. Arm B subjects will continue to receive the anti-HER2 therapy. It is expected that the addition of palbociclib to the first-line treatment of HER2 disease will delay the onset of therapeutic resistance and ultimately prolong the survival of patients with metastatic breast cancer. The study is designed to treat the subset of patients with HER2+ disease who are also hormone receptor positive (HR+). It is also expected that palbociclib will modulate the endocrine resistance in HER2+/HR+ disease and potentiate the benefits of anti-HER2 therapy. Lastly, the current study includes a comprehensive molecular characterization of the disease at study entrance which will allow us to investigate the benefits of palbociclib in subsets of HER2+/HR+ disease such as PIK3CA mutant.

ELIGIBILITY:
Inclusion Criteria (Preliminary Screening)

1. Signed Preliminary Screening Informed Consent Form obtained prior to any study specific assessments and procedures
2. Age ≥18 years (or per national guidelines)
3. Patients must have histologically confirmed invasive breast cancer that is metastatic or not amenable for resection or radiation therapy with curative intent. Histological documentation of metastatic/recurrent breast cancer is not required if there is unequivocal evidence for recurrence of the breast cancer.
4. Patients must have histologically confirmed HER2+ and hormone receptor positive (ER+ and/or PR+), metastatic breast cancer. ER, PR and HER2 measurements should be performed according to institutional guidelines, in a CLIA-approved setting in the US or certified laboratories for Non-US regions. Cut-off values for positive/negative staining should be in accordance with current ASCO/CAP (American Society of Clinical Oncology/College of American Pathologists) guidelines.
5. Patients must agree to provide a representative formalin-fixed paraffin-embedded (FFPE) tumor tissue block (preferred) from primary breast or metastatic site (archival) OR at least 15 freshly cut unstained slides from such a block, along with a pathology report documenting HER2 positivity and hormone receptor positivity.
6. Patients should be willing to provide a representative tumor specimen obtained from recently biopsied metastatic disease if clinically feasible. This is recommended but optional tissue.

   Inclusion Criteria (Randomization Screening)
7. Signed Main Informed Consent Form obtained prior to any study specific assessments and procedures
8. Age ≥ 18 years (or per national guidelines)
9. ECOG performance status 0-1
10. Patients must be able and willing to swallow and retain oral medication without a condition that would interfere with enteric absorption.
11. Serum or urine pregnancy test must be negative within 7 days of randomization in women of childbearing potential. Pregnancy testing does not need to be pursued in patients who are judged as postmenopausal before randomization, as determined by local practice, or who have undergone bilateral oophorectomy, total hysterectomy, or bilateral tubal ligation. Women of childbearing potential and male patients randomized into the study must use adequate contraception for the duration of protocol treatment which is 6 months after the last treatment with palbociclib if they are in Arm A and for 7 months after last treatment with trastuzumab if in either Arm A or Arm B Adequate contraception is defined as one highly effective form (i.e. abstinence, (fe)male sterilization OR two effective forms (e.g. non-hormonal IUD and condom / occlusive cap with spermicidal foam / gel / film / cream / suppository).
12. Resolution of all acute toxic effects of prior induction anti-HER2-based chemotherapy regimen to NCI CTCAE version 4.0 Grade ≤1 (except alopecia or other toxicities not considered a safety risk for the patient at investigator's discretion) 12 weeks between last dose of chemotherapy-anti-HER2therapy and randomization are allowed. Endocrine therapy could start before study randomization.
13. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures

    Prior Treatment Specifics
14. Patients may or may not have received neo/adjuvant therapy, but must have a disease-free interval from completion of anti-HER2 therapy to metastatic diagnosis ≥6 months.
15. Patients must have received an acceptable, standard, chemotherapy containing anti-HER2 based induction therapy for the treatment of metastatic breast cancer prior to study enrollment. For this study, chemotherapy is limited to a taxane or vinorelbine (only for trastuzumab-based regimen). Eligible patients are expected to have completed 6 cycles of chemotherapy containing anti-HER2-therapy treatment. A minimum of 4 cycles of treatment is acceptable for patients experiencing significant toxicity associated with treatment as long as they are without evidence of disease progression (i.e. CR, PR or SD). The maximum number of cycles is 8. Patients can randomize immediately following completion of their induction therapy, or for those who have already completed induction, a gap of 12 weeks between their last infusion/dose of induction therapy and the C1D1 visit is permitted. Patients are eligible provided they are without evidence of disease progression by local assessment (i.e. CR, PR or SD).
16. Patients with a history or presence of asymptomatic CNS metastases are eligible, provided they meet all of the following criteria:

    * Disease outside the CNS is present.
    * No evidence of interim progression between the completion of induction therapy and the screening radiographic study
    * No history of intracranial hemorrhage or spinal cord hemorrhage
    * Not requiring anti-convulsants for symptomatic control
    * Minimum of 3 weeks between completion of CNS radiotherapy and Cycle 1 Day 1 and recovery from significant (Grade ≥ 3) acute toxicity with no ongoing requirement for corticosteroid

    Baseline Body Function Specifics
17. Absolute neutrophil count ≥ 1,000/mm3
18. Platelets ≥ 100,000/mm3
19. Hemoglobin ≥ 10g/dL
20. Total serum bilirubin ≤ ULN; or total bilirubin ≤ 3.0 × ULN with direct bilirubin within normal range in patients with documented Gilbert's Syndrome.
21. Aspartate aminotransferase (AST or SGOT) and alanine aminotransferase (ALT or SGPT) ≤ 3 × institutional ULN (≤5 x ULN if liver metastases are present).
22. Serum creatinine below the upper limit of normal (ULN) of the institutional normal range or creatinine clearance ≥ 60 mL/min/1.73 m2 for patients with serum creatinine levels above institutional ULN.
23. Left ventricular ejection fraction (LVEF) ≥ 50% at baseline as determined by either ECHO or MUGA

Exclusion Criteria (Randomization)

1. Concurrent therapy with other Investigational Products.
2. Prior therapy with any CDK 4/6 inhibitor.
3. History of allergic reactions attributed to compounds of chemical or biologic composition similar to palbociclib.
4. Patients receiving any medications or substances that are strong inhibitors or inducers of CYP3A isoenzymes within 7 days of randomization (see Section 8.6.3 for list of strong inhibitors or inducers of CYP3A isoenzymes).
5. Uncontrolled current illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, diabetes, or psychiatric illness/social situations that would limit compliance with study requirements. Ability to comply with study requirements is to be assessed by each investigator at the time of screening for study participation.
6. Pregnant women, or women of childbearing potential without a negative pregnancy test (serum or urine) within 7 days prior to randomization, irrespective of the method of contraception used, are excluded from this study because the effect of palbociclib on a developing fetus is unknown. Breastfeeding must be discontinued prior to study entry.
7. Patients on combination antiretroviral therapy, i.e. those who are HIV-positive, are ineligible because of the potential for pharmacokinetic interactions or increased immunosuppression with palbociclib.
8. QTc interval >480 msec, Brugada syndrome or known history of QTc prolongation or Torsade de Pointes.
9. Patients with clinically significant history of liver disease, including viral or other known hepatitis, current alcohol abuse, or cirrhosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 518 (Actual)
Dates: Start 2017-06-21 (Actual); Primary Completion 2024-10-15 (Actual); Study Completion 2026-07-31 (Estimated)

CONTACTS AND LOCATIONS:
Locations (106):
- United States (35):
  - UCSF, San Francisco, California
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Baycare Healthcare (Morton Plant Mease), Clearwater, Florida
  - Memorial Healthcare System, Hollywood, Florida
  - University of Miami, Miami, Florida
  - Florida Hospital, Orlando, Florida
  - Emory University, Atlanta, Georgia
  - University of Illinois at Chicago, Chicago, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - Cancer Center of Kansas, Wichita, Kansas
  - Ochsner Medical Center Jefferson, New Orleans, Louisiana
  - New England Cancer Specialists, Scarborough, Maine
  - University of Maryland - Greenebaum Comprehensive Cancer Center, Baltimore, Maryland
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Lowell General Hospital, Lowell, Massachusetts
  - Michigan Cancer Research Consortium (St. Joseph Mercy Hospital, Ann Arbor, Michigan
  - West Michigan Cancer Center, Grand Rapids, Michigan
  - Metro-Minnesota NCI Community Oncology Research Program, Minneapolis, Minnesota
  - Mayo Clinic, Rochester, MN, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Nebraska Methodist Hospital, Omaha, Nebraska
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Hackensack Medical Center, Hackensack, New Jersey
  - The Valley Hospital, Okonite Research Center, Paramus, New Jersey
  - New Mexico Cancer Care Alliance, Albuquerque, New Mexico
  - Duke Cancer Institute, Durham, North Carolina
  - First Health of the Carolinas Cancer Center, Pinehurst, North Carolina
  - Ohio State University, Columbus, Ohio
  - Legacy Good Samaritan Hospital, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Lexington Medical Center, West Columbia, South Carolina
  - Vanderbilt University Medical Center, Nashville, Tennessee
  - MD Anderson, Houston, Texas
  - Huntsman Cancer Institute, University of Utah, Salt Lake City, Utah
- Australia (9):
  - Monash Health, Clayton
  - St. Vincent's Hospital, Sydney Kinghorn Cancer Centre, Darlinghurst
  - The Canberra Hospital, Garran
  - Peter MacCallum Cancer Centre, Royal Melbourne Hospital, Melbourne
  - Breast Cancer Research Centre-WA, Nedlands
  - Icon Cancer Care, South Brisbane
  - Mater Cancer Care Centre, South Brisbane
  - Calvary Mater Newcastle Hospital, Waratah
  - Westmead Hospital, Westmead
- France (25):
  - Institut de Cancérologie de l'Ouest, site Paul Papin, Angers
  - Institut Sainte Catherine, Avignon
  - Institut Bergonié, Bordeaux
  - Centre Francois Baclesse, Caen
  - Centre Hospitalier Cholet, Cholet
  - Centre Jean Perrin, Clermont-Ferrand
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - CHU de Limoges, Limoges
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - Institut de Cancerologie de Montpellier, Montpellier
  - Centre Azureen de Cancerologie, Mougins
  - Centre Antoine Lacassagne, Nice
  - Institut Curie Site Paris, Paris
  - Tenon Oncologie Médicale - APHP, Paris
  - Centre CARIO-HPCA, Plérin
  - Institut Jean Godinot, Reims
  - Centre Eugene Marquis, Rennes
  - Centre Henri Becquerel, Rouen
  - Institut Curie Site Saint Cloud, Saint-Cloud
  - Institut de Cancérologie Lucien Neuwirth, Saint-Priest-en-Jarez
  - Centre Paul Strauss, Strasbourg
  - Intitut Claudius Regaud, Toulouse
  - Gustave Roussy, Villejuif
- Germany (9):
  - Marienhospital Bottrop, Bottrop
  - St. Elisabeth Krankenhaus, Cologne
  - Kliniken Essen-Mitte, Evang. Huyssens-Stiftung/Knappschaft GmbH, Essen
  - Agaplesion Markus Krankenhaus, Frankfurt
  - Diakovere Henriettenstift Frauenklinik, Hanover
  - UKSH, Klinik für Gynäkologie und Geburtshilfe, Kiel
  - Praxis Prof. Nitz im Brustzentrum Niederrhein, Münster
  - Universitätsklinikum Münster, Münster
  - Leopoldina-Krankenhaus Schweinfurt, Schweinfurt
- Italy (5):
  - Policlinico Sant'Orsola-Malpighi, Bologna
  - U.O. Oncologia AOU Arcispedale Sant'Anna, Cona
  - Istituto Europeo di Oncologia, Milan
  - Ospedale San Raffaele, Segrate
  - Ospedale Santa Maria della Misericordia, Udine
- Auckland City Hospital Cancer and Blood Research, Auckland, New Zealand
- Portugal (4):
  - Hospital Champalimaud, Lisbon
  - Hospital Da Luz, Lisbon
  - Hospital Beatriz Angelo, Loures
  - IPO Porto, Porto
- Spain (18):
  - Hospital Clínic de Barcelona, Barcelona
  - Hospital General de Catalunya, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - ICO L'Hospitalet, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid
  - Hospital Universitario de Fuenlabrada, Madrid
  - Hospital Universitario Fundación Alcorcón, Madrid
  - Hospital Universitario Fundación Jiménez Díaz, Madrid
  - Hospital Universitario La Paz, Madrid
  - MD Anderson Cancer Center Spain, Madrid
  - Hospital Regional Universitario de Málaga, Málaga
  - Hospital Universitario Virgen de la Arrixaca, Murcia
  - Complejo Hospitalario de Navarra, Navarro
  - Hospital Universitario de Salamanca, Salamanca
  - Complejo Hospitalario Univ. De Santiago, Santiago
  - Hospital Quirón Sagrado Corazón, Seville
  - Hospital Sant Joan de Reus, Tarragona
  - Hospital Clínico Universitario de Valencia, Valencia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Early Breast Cancer Trialists' Collaborative Group (EBCTCG); Peto R, Davies C, Godwin J, Gray R, Pan HC, Clarke M, Cutter D, Darby S, McGale P, Taylor C, Wang YC, Bergh J, Di Leo A, Albain K, Swain S, Piccart M, Pritchard K. Comparisons between different polychemotherapy regimens for early breast cancer: meta-analyses of long-term outcome among 100,000 women in 123 randomised trials. Lancet. 2012 Feb 4;379(9814):432-44. doi: 10.1016/S0140-6736(11)61625-5. Epub 2011 Dec 5. PMID 22152853
- [Background] Welch HG, Gorski DH, Albertsen PC. Trends in Metastatic Breast and Prostate Cancer--Lessons in Cancer Dynamics. N Engl J Med. 2015 Oct 29;373(18):1685-7. doi: 10.1056/NEJMp1510443. No abstract available. PMID 26510017
- [Background] Baselga J, Cortes J, Kim SB, Im SA, Hegg R, Im YH, Roman L, Pedrini JL, Pienkowski T, Knott A, Clark E, Benyunes MC, Ross G, Swain SM; CLEOPATRA Study Group. Pertuzumab plus trastuzumab plus docetaxel for metastatic breast cancer. N Engl J Med. 2012 Jan 12;366(2):109-19. doi: 10.1056/NEJMoa1113216. Epub 2011 Dec 7. PMID 22149875
- [Background] Swain SM, Baselga J, Kim SB, Ro J, Semiglazov V, Campone M, Ciruelos E, Ferrero JM, Schneeweiss A, Heeson S, Clark E, Ross G, Benyunes MC, Cortes J; CLEOPATRA Study Group. Pertuzumab, trastuzumab, and docetaxel in HER2-positive metastatic breast cancer. N Engl J Med. 2015 Feb 19;372(8):724-34. doi: 10.1056/NEJMoa1413513. PMID 25693012
- [Background] Ferlay J, Steliarova-Foucher E, Lortet-Tieulent J, Rosso S, Coebergh JW, Comber H, Forman D, Bray F. Cancer incidence and mortality patterns in Europe: estimates for 40 countries in 2012. Eur J Cancer. 2013 Apr;49(6):1374-403. doi: 10.1016/j.ejca.2012.12.027. Epub 2013 Feb 26. PMID 23485231
- [Background] Sherr CJ, Roberts JM. CDK inhibitors: positive and negative regulators of G1-phase progression. Genes Dev. 1999 Jun 15;13(12):1501-12. doi: 10.1101/gad.13.12.1501. No abstract available. PMID 10385618
- [Background] van den Heuvel S, Harlow E. Distinct roles for cyclin-dependent kinases in cell cycle control. Science. 1993 Dec 24;262(5142):2050-4. doi: 10.1126/science.8266103.
- [Background] Weinberg RA. The retinoblastoma protein and cell cycle control. Cell. 1995 May 5;81(3):323-30. doi: 10.1016/0092-8674(95)90385-2. No abstract available. PMID 7736585
- [Background] Harper JW, Adami GR, Wei N, Keyomarsi K, Elledge SJ. The p21 Cdk-interacting protein Cip1 is a potent inhibitor of G1 cyclin-dependent kinases. Cell. 1993 Nov 19;75(4):805-16. doi: 10.1016/0092-8674(93)90499-g. PMID 8242751
- [Background] Koff A, Ohtsuki M, Polyak K, Roberts JM, Massague J. Negative regulation of G1 in mammalian cells: inhibition of cyclin E-dependent kinase by TGF-beta. Science. 1993 Apr 23;260(5107):536-9. doi: 10.1126/science.8475385.
- [Background] Polyak K, Kato JY, Solomon MJ, Sherr CJ, Massague J, Roberts JM, Koff A. p27Kip1, a cyclin-Cdk inhibitor, links transforming growth factor-beta and contact inhibition to cell cycle arrest. Genes Dev. 1994 Jan;8(1):9-22. doi: 10.1101/gad.8.1.9. PMID 8288131
- [Background] Sherr CJ. D-type cyclins. Trends Biochem Sci. 1995 May;20(5):187-90. doi: 10.1016/s0968-0004(00)89005-2. PMID 7610482
- [Background] Toyoshima H, Hunter T. p27, a novel inhibitor of G1 cyclin-Cdk protein kinase activity, is related to p21. Cell. 1994 Jul 15;78(1):67-74. doi: 10.1016/0092-8674(94)90573-8. PMID 8033213
- [Background] Lukas J, Parry D, Aagaard L, Mann DJ, Bartkova J, Strauss M, Peters G, Bartek J. Retinoblastoma-protein-dependent cell-cycle inhibition by the tumour suppressor p16. Nature. 1995 Jun 8;375(6531):503-6. doi: 10.1038/375503a0. PMID 7777060
- [Background] Medema RH, Herrera RE, Lam F, Weinberg RA. Growth suppression by p16ink4 requires functional retinoblastoma protein. Proc Natl Acad Sci U S A. 1995 Jul 3;92(14):6289-93. doi: 10.1073/pnas.92.14.6289. PMID 7603984
- [Background] Lee RJ, Albanese C, Fu M, D'Amico M, Lin B, Watanabe G, Haines GK 3rd, Siegel PM, Hung MC, Yarden Y, Horowitz JM, Muller WJ, Pestell RG. Cyclin D1 is required for transformation by activated Neu and is induced through an E2F-dependent signaling pathway. Mol Cell Biol. 2000 Jan;20(2):672-83. doi: 10.1128/MCB.20.2.672-683.2000. PMID 10611246
- [Background] Lane HA, Beuvink I, Motoyama AB, Daly JM, Neve RM, Hynes NE. ErbB2 potentiates breast tumor proliferation through modulation of p27(Kip1)-Cdk2 complex formation: receptor overexpression does not determine growth dependency. Mol Cell Biol. 2000 May;20(9):3210-23. doi: 10.1128/MCB.20.9.3210-3223.2000. PMID 10757805
- [Background] Yu Q, Sicinska E, Geng Y, Ahnstrom M, Zagozdzon A, Kong Y, Gardner H, Kiyokawa H, Harris LN, Stal O, Sicinski P. Requirement for CDK4 kinase function in breast cancer. Cancer Cell. 2006 Jan;9(1):23-32. doi: 10.1016/j.ccr.2005.12.012. PMID 16413469
- [Background] Nahta R, Iglehart JD, Kempkes B, Schmidt EV. Rate-limiting effects of Cyclin D1 in transformation by ErbB2 predicts synergy between herceptin and flavopiridol. Cancer Res. 2002 Apr 15;62(8):2267-71. PMID 11956082
- [Background] Reddy HK, Mettus RV, Rane SG, Grana X, Litvin J, Reddy EP. Cyclin-dependent kinase 4 expression is essential for neu-induced breast tumorigenesis. Cancer Res. 2005 Nov 15;65(22):10174-8. doi: 10.1158/0008-5472.CAN-05-2639. PMID 16288002
- [Background] Yang C, Ionescu-Tiba V, Burns K, Gadd M, Zukerberg L, Louis DN, Sgroi D, Schmidt EV. The role of the cyclin D1-dependent kinases in ErbB2-mediated breast cancer. Am J Pathol. 2004 Mar;164(3):1031-8. doi: 10.1016/S0002-9440(10)63190-2. PMID 14982856
- [Background] Landis MW, Pawlyk BS, Li T, Sicinski P, Hinds PW. Cyclin D1-dependent kinase activity in murine development and mammary tumorigenesis. Cancer Cell. 2006 Jan;9(1):13-22. doi: 10.1016/j.ccr.2005.12.019. PMID 16413468
- [Background] Finn RS, Dering J, Conklin D, Kalous O, Cohen DJ, Desai AJ, Ginther C, Atefi M, Chen I, Fowst C, Los G, Slamon DJ. PD 0332991, a selective cyclin D kinase 4/6 inhibitor, preferentially inhibits proliferation of luminal estrogen receptor-positive human breast cancer cell lines in vitro. Breast Cancer Res. 2009;11(5):R77. doi: 10.1186/bcr2419. PMID 19874578
- [Background] Witkiewicz AK, Cox DW, Rivadeneira D, Ertel AE, Fortina P, Schwartz GF, Knudsen ES. The retinoblastoma tumor suppressor pathway modulates the invasiveness of ErbB2-positive breast cancer. Oncogene. 2014 Jul 24;33(30):3980-91. doi: 10.1038/onc.2013.367. Epub 2013 Oct 14. PMID 24121271
- [Background] Roberts PJ, Bisi JE, Strum JC, Combest AJ, Darr DB, Usary JE, Zamboni WC, Wong KK, Perou CM, Sharpless NE. Multiple roles of cyclin-dependent kinase 4/6 inhibitors in cancer therapy. J Natl Cancer Inst. 2012 Mar 21;104(6):476-87. doi: 10.1093/jnci/djs002. Epub 2012 Feb 1. PMID 22302033
- [Background] Goel S, Wang Q, Watt AC, Tolaney SM, Dillon DA, Li W, Ramm S, Palmer AC, Yuzugullu H, Varadan V, Tuck D, Harris LN, Wong KK, Liu XS, Sicinski P, Winer EP, Krop IE, Zhao JJ. Overcoming Therapeutic Resistance in HER2-Positive Breast Cancers with CDK4/6 Inhibitors. Cancer Cell. 2016 Mar 14;29(3):255-269. doi: 10.1016/j.ccell.2016.02.006. PMID 26977878
- [Background] Cristofanilli M, Turner NC, Bondarenko I, Ro J, Im SA, Masuda N, Colleoni M, DeMichele A, Loi S, Verma S, Iwata H, Harbeck N, Zhang K, Theall KP, Jiang Y, Bartlett CH, Koehler M, Slamon D. Fulvestrant plus palbociclib versus fulvestrant plus placebo for treatment of hormone-receptor-positive, HER2-negative metastatic breast cancer that progressed on previous endocrine therapy (PALOMA-3): final analysis of the multicentre, double-blind, phase 3 randomised controlled trial. Lancet Oncol. 2016 Apr;17(4):425-439. doi: 10.1016/S1470-2045(15)00613-0. Epub 2016 Mar 3. PMID 26947331
- [Background] Ramakrishna N, Temin S, Chandarlapaty S, Crews JR, Davidson NE, Esteva FJ, Giordano SH, Gonzalez-Angulo AM, Kirshner JJ, Krop I, Levinson J, Modi S, Patt DA, Perez EA, Perlmutter J, Winer EP, Lin NU. Recommendations on disease management for patients with advanced human epidermal growth factor receptor 2-positive breast cancer and brain metastases: American Society of Clinical Oncology clinical practice guideline. J Clin Oncol. 2014 Jul 1;32(19):2100-8. doi: 10.1200/JCO.2013.54.0955. Epub 2014 May 5. PMID 24799487
- [Background] Cardoso F, Costa A, Norton L, Senkus E, Aapro M, Andre F, Barrios CH, Bergh J, Biganzoli L, Blackwell KL, Cardoso MJ, Cufer T, El Saghir N, Fallowfield L, Fenech D, Francis P, Gelmon K, Giordano SH, Gligorov J, Goldhirsch A, Harbeck N, Houssami N, Hudis C, Kaufman B, Krop I, Kyriakides S, Lin UN, Mayer M, Merjaver SD, Nordstrom EB, Pagani O, Partridge A, Penault-Llorca F, Piccart MJ, Rugo H, Sledge G, Thomssen C, Van't Veer L, Vorobiof D, Vrieling C, West N, Xu B, Winer E. ESO-ESMO 2nd international consensus guidelines for advanced breast cancer (ABC2)dagger. Ann Oncol. 2014 Oct;25(10):1871-1888. doi: 10.1093/annonc/mdu385. Epub 2014 Sep 18. No abstract available. PMID 25234545
- [Background] Lipton A, Ali SM, Leitzel K, Demers L, Harvey HA, Chaudri-Ross HA, Brady C, Wyld P, Carney W. Serum HER-2/neu and response to the aromatase inhibitor letrozole versus tamoxifen. J Clin Oncol. 2003 May 15;21(10):1967-72. doi: 10.1200/JCO.2003.09.098. PMID 12743150
- [Background] Burstein HJ, Harris LN, Marcom PK, Lambert-Falls R, Havlin K, Overmoyer B, Friedlander RJ Jr, Gargiulo J, Strenger R, Vogel CL, Ryan PD, Ellis MJ, Nunes RA, Bunnell CA, Campos SM, Hallor M, Gelman R, Winer EP. Trastuzumab and vinorelbine as first-line therapy for HER2-overexpressing metastatic breast cancer: multicenter phase II trial with clinical outcomes, analysis of serum tumor markers as predictive factors, and cardiac surveillance algorithm. J Clin Oncol. 2003 Aug 1;21(15):2889-95. doi: 10.1200/JCO.2003.02.018. PMID 12885806
- [Background] Chan A, Martin M, Untch M, Gil MG, Guillem-Porta V, Wojtukiewicz M, Kellokumpu-Lehtinen P, Sommer HL, Georgoulias V, Battelli N, Pawlicki M, Aubert D, Bourlard T, Gasmi J, Villanova G, Petruzelka L; Navelbine Herceptin Project. Vinorelbine plus trastuzumab combination as first-line therapy for HER 2-positive metastatic breast cancer patients: an international phase II trial. Br J Cancer. 2006 Oct 9;95(7):788-93. doi: 10.1038/sj.bjc.6603351. Epub 2006 Sep 12. PMID 16969343
- [Background] Brady MJ, Cella DF, Mo F, Bonomi AE, Tulsky DS, Lloyd SR, Deasy S, Cobleigh M, Shiomoto G. Reliability and validity of the Functional Assessment of Cancer Therapy-Breast quality-of-life instrument. J Clin Oncol. 1997 Mar;15(3):974-86. doi: 10.1200/JCO.1997.15.3.974. PMID 9060536
- [Background] EuroQol Group. EuroQol--a new facility for the measurement of health-related quality of life. Health Policy. 1990 Dec;16(3):199-208. doi: 10.1016/0168-8510(90)90421-9. PMID 10109801
- [Result] Finn RS, Crown JP, Lang I, Boer K, Bondarenko IM, Kulyk SO, Ettl J, Patel R, Pinter T, Schmidt M, Shparyk Y, Thummala AR, Voytko NL, Fowst C, Huang X, Kim ST, Randolph S, Slamon DJ. The cyclin-dependent kinase 4/6 inhibitor palbociclib in combination with letrozole versus letrozole alone as first-line treatment of oestrogen receptor-positive, HER2-negative, advanced breast cancer (PALOMA-1/TRIO-18): a randomised phase 2 study. Lancet Oncol. 2015 Jan;16(1):25-35. doi: 10.1016/S1470-2045(14)71159-3. Epub 2014 Dec 16. PMID 25524798
- [Result] Finn, R.S., et al., PALOMA-2: Primary results from a phase III trial of palbociclib (P) with letrozole (L) compared with letrozole alone in postmenopausal women with ER+/HER2- advanced breast cancer (ABC). ASCO Meeting Abstracts, 2016. 34(15_suppl): p. 507.
- [Result] Paridaens R, Dirix L, Lohrisch C, Beex L, Nooij M, Cameron D, Biganzoli L, Cufer T, Duchateau L, Hamilton A, Lobelle JP, Piccart M; European Organization for the Research and Treatment of Cancer (EORTC)- Investigational Drug Branch for Breast Cancer (IDBBC). Mature results of a randomized phase II multicenter study of exemestane versus tamoxifen as first-line hormone therapy for postmenopausal women with metastatic breast cancer. Ann Oncol. 2003 Sep;14(9):1391-8. doi: 10.1093/annonc/mdg362. PMID 12954578
- [Result] Pfizer, Inc. Palbociclib (PD-0332991): Investigator's Brochure. N.p.: Pfizer, 2015. Print.
- [Derived] Metzger O, Mandrekar S, Goel S, Gligorov J, Lim E, Ciruelos E, Loibl S, Dockter T, Gonzalez Farre X, Francis PA, Lynce F, Lanzillotti J, DuFrane C, Wall A, Strand C, Krop I, Vaz-Luis I, Tripathy D, Loi S, Prat A, Goetz M, Escriva-de-Romani S, Porter D, Spoenlein J, Stover DG, Sardesai S, Heudel P, Koehler M, Huang Bartlett C, Holynskyj A, Gopalakrishna P, Gauthier E, Delaloge S, Miller K, Winer EP, Gianni L, Partridge AH, DeMichele A, Carey LA. Palbociclib for Hormone-Receptor-Positive, HER2-Positive Advanced Breast Cancer. N Engl J Med. 2026 Jan 29;394(5):451-462. doi: 10.1056/NEJMoa2511218. PMID 41604639
- [Derived] Peddi PF, Slamon DJ. Frontiers in HER2-positive breast cancer in 2020. Curr Opin Obstet Gynecol. 2021 Feb 1;33(1):48-52. doi: 10.1097/GCO.0000000000000677. PMID 33369581

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm A: Palbociclib 125 mg daily and AntiHER2 Therapy (trastuzumab/pertuzumab) q3wks + Endocrine Therapy (letrozole, anastrozole, exemstane OR fulvestratnt)
- Arm B: AntiHER2 Therapy (trastuzumab/pertuzumab) q3wks + Endocrine Therapy (letrozole, anastrozole, exemstane OR fulvestrant)
Period: Overall Study
Arm/Group | Arm A | Arm B
Started | 261 | 257
Completed | 261 | 257
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A | Arm B | Total
Number analyzed (Participants) | 261 | 257 | 518
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 53.5 [43.6 to 60.4] | 53 [45.1 to 62.8] | 53.4 [44.2 to 61.4]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 259 | 256 | 515
  Male | 2 | 1 | 3
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 46 | 25 | 71
  Not Hispanic or Latino | 120 | 136 | 256
  Unknown or Not Reported | 95 | 96 | 191
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 8 | 3 | 11
  Native Hawaiian or Other Pacific Islander | 3 | 3 | 6
  Black or African American | 4 | 11 | 15
  White | 207 | 194 | 401
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 36 | 45 | 81

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) as Assessed by Investigator
Description: The time from registration to disease progression or death.
Time Frame: 7 years 3 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 261 | 257
months | 44.3 [32.4 to 56.8] | 29.1 [23.3 to 38.6]

2. Secondary Outcome: Overall Survival (OS)
Description: Defined as time from date of randomization to date of death due to any cause
Time Frame: 7 years 3 months
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 261 | 257
Months | NA [71.6 to NA] — Too few events occurred to calculate the median and upper CI limit | 77 [72 to NA] — Too few events occurred to calculate the upper CI limit

3. Secondary Outcome: 3 and 5 Year Survival Probabilities
Description: Defined as the percentage of patients still alive and followed at 3 and 5 years post beginning of treatment.
Time Frame: 5 years
Measure: Number (95% Confidence Interval); unit: percentage of patients alive
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 261 | 257
percentage of patients alive
  At 3 years | 87 [82.8 to 91.2] | 84.7 [80 to 89.3]
  At 5 years | 72.9 [66 to 79.7] | 68.5 [61.1 to 76]

4. Secondary Outcome: Objective Response Rate (OR: CR or PR)
Description: Defined as proportion of patients that achieve complete response (CR) or partial response (PR) according to RECIST v1.1. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.1) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 24 months
Population: Patients evaluated for disease
Measure: Number; unit: proportion of participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 231 | 230
proportion of participants | 0.329 | 0.248

5. Secondary Outcome: Duration of Response (DOR)
Description: Defined as the time from the first documentation of objective tumor response (CR or PR) to the first documentation of objective tumor progression or to death from any cause, whichever occurs first
Time Frame: 72 months
Population: Patients that achieved confirmed response
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 76 | 57
Months | 44.9 [27.1 to 51.6] | 30.8 [26.0 to NA] — Upper limit not available due to low number of events

6. Secondary Outcome: Clinical Benefit Rate
Description: The Clinical Benefit Rate (CBR) on each treatment arm will be estimated by dividing the number of patients with CR, PR, or SD/Non-CR and Non-PD (for patients with measurable disease) for ≥ 24 weeks by the number of patients randomized to the treatment arm.
Time Frame: 24 months
Measure: Number; unit: proportion of participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 261 | 257
proportion of participants | 0.889 | 0.809

7. Secondary Outcome: Incidence of Grade 3 or Higher Adverse Events (as Graded by NCI CTCAE v 4.0)
Description: The proportion of patient by arm that experienced grade 3 or higher adverse events will be reported
Time Frame: 24 months
Measure: Number; unit: proportion of participants
Arm/Group | Arm A | Arm B
Number analyzed (Participants) | 261 | 257
proportion of participants | 0.797 | 0.306

8. Secondary Outcome: Patient Reported Outcomes
Description: Time to symptom progression (FACT-B PFB-TOI), breast cancer specific health treatment related quality of life and general health status
Time Frame: 24 months
Reporting Status: Not Posted

9. Secondary Outcome: Incidence of CNS Metastasis
Description: Compare the incidence of CNS metastasis between treatment arms
Time Frame: 24 months
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Trough Plasma Concentration of Palbociclib, Trastuzumab and Pertuzumab
Description: only for patients enrolled in the US
Time Frame: Palbociclib PK assessment: Day 22, Cycle 1, No; Pertuzumab, Trastuzumab PK assessment: Day 1, Cycle 4
Reporting Status: Not Posted

11. Other Pre Specified Outcome: PIK3CA Genotype Assessed in Circulating cfDNA
Description: Progression Free Survival (PFS) based upon investigator assessment of progression between patients in the two treatment arms in the subset of patients with tumors bearing a PIK3CA mutation.
Time Frame: Day 1, Cycle 1, Day 1, Cycle 4, End of Treatment, approx 24 months
Reporting Status: Not Posted

12. Other Pre Specified Outcome: Tumor Tissue Biomarkers Including Genes, Proteins, and RNA Expression
Description: Will evaluate baseline tumor and blood-based markers as predictors of benefit from the addition of palbociclib to anti-HER2 therapy plus endocrine therapy
Time Frame: Baseline
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 5 years for adverse events and 7 years 3 months for mortality
Arm/Group | Arm A | Arm B
All-Cause Mortality (participants affected / at risk) | 60/261 | 63/257
Serious Adverse Events (participants affected / at risk) | 75/261 | 54/257
Other Adverse Events (participants affected / at risk) | 261/261 | 234/257
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=261) | Arm B (N=257)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 0 (0) | 1 (1)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 3 (3) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Heart failure (Cardiac disorders) | 0 (0) | 1 (1)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Pericardial effusion (Cardiac disorders) | 0 (0) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Endocrine disorders - Other, specify (Endocrine disorders) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 0 (0) | 1 (1)
Eye disorders - Other, specify (Eye disorders) | 0 (0) | 1 (1)
Papilledema (Eye disorders) | 0 (0) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 4 (4) | 2 (2)
Anal fistula (Gastrointestinal disorders) | 1 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colonic hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Gastric ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 4 (5) | 1 (1)
Gastrointestinal pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Jejunal perforation (Gastrointestinal disorders) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 2 (2) | 0 (0)
Pancreatitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 4 (4) | 1 (2)
Vomiting (Gastrointestinal disorders) | 2 (2) | 1 (1)
Death NOS (General disorders) | 4 (4) | 4 (4)
Fever (General disorders) | 4 (4) | 0 (0)
Flu like symptoms (General disorders) | 1 (1) | 0 (0)
Gen disord and admin site conds-Oth spec (General disorders) | 1 (1) | 5 (5)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Pain (General disorders) | 3 (3) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 4 (4) | 2 (2)
Hepatic hemorrhage (Hepatobiliary disorders) | 1 (1) | 0 (0)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 0 (0) | 1 (1)
Abdominal infection (Infections and infestations) | 0 (0) | 1 (1)
Appendicitis (Infections and infestations) | 0 (0) | 1 (1)
Bronchial infection (Infections and infestations) | 1 (1) | 0 (0)
Catheter related infection (Infections and infestations) | 0 (0) | 2 (2)
Device related infection (Infections and infestations) | 0 (0) | 1 (2)
Duodenal infection (Infections and infestations) | 1 (1) | 0 (0)
Endocarditis infective (Infections and infestations) | 1 (1) | 0 (0)
Enterocolitis infectious (Infections and infestations) | 0 (0) | 1 (1)
Infections and infestations - Oth spec (Infections and infestations) | 10 (11) | 4 (5)
Joint infection (Infections and infestations) | 0 (0) | 1 (1)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1)
Lung infection (Infections and infestations) | 3 (3) | 2 (2)
Sepsis (Infections and infestations) | 3 (3) | 1 (1)
Skin infection (Infections and infestations) | 1 (1) | 0 (0)
Small intestine infection (Infections and infestations) | 1 (1) | 0 (0)
Upper respiratory infection (Infections and infestations) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 5 (5) | 2 (2)
Aortic injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fracture (Injury, poisoning and procedural complications) | 6 (6) | 3 (3)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Dehydration (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 2 (2)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3 (4) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 0 (0) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1) | 1 (1)
Headache (Nervous system disorders) | 4 (4) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1)
Nervous system disorders - Oth spec (Nervous system disorders) | 3 (5) | 1 (1)
Peripheral motor neuropathy (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 2 (2) | 1 (1)
Stroke (Nervous system disorders) | 1 (1) | 1 (1)
Syncope (Nervous system disorders) | 1 (1) | 3 (3)
Transient ischemic attacks (Nervous system disorders) | 1 (1) | 0 (0)
Confusion (Psychiatric disorders) | 1 (2) | 0 (0)
Delirium (Psychiatric disorders) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 2 (2) | 1 (1)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 1 (2) | 0 (0)
Renal colic (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 4 (5)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 4 (6)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Surgical and medical proced - Oth spec (Surgical and medical procedures) | 0 (0) | 1 (1)
Hematoma (Vascular disorders) | 1 (1) | 0 (0)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Thromboembolic event (Vascular disorders) | 1 (1) | 1 (1)
Vascular disorders - Other, specify (Vascular disorders) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A (N=261) | Arm B (N=257)
Anemia (Blood and lymphatic system disorders) | 84 (205) | 24 (75)
Blood and lymph sys disorders - Oth Spec (Blood and lymphatic system disorders) | 21 (38) | 8 (13)
Bone marrow hypocellular (Blood and lymphatic system disorders) | 3 (4) | 0 (0)
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Hemolysis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Leukocytosis (Blood and lymphatic system disorders) | 2 (2) | 1 (1)
Lymph node pain (Blood and lymphatic system disorders) | 2 (2) | 2 (2)
Thrombotic thrombocytopenic purpura (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Aortic valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Cardiac disorders - Other, specify (Cardiac disorders) | 8 (8) | 2 (2)
Chest pain - cardiac (Cardiac disorders) | 0 (0) | 2 (2)
Heart failure (Cardiac disorders) | 0 (0) | 2 (3)
Left ventricular systolic dysfunction (Cardiac disorders) | 0 (0) | 1 (1)
Mitral valve disease (Cardiac disorders) | 2 (2) | 1 (1)
Palpitations (Cardiac disorders) | 3 (4) | 5 (5)
Pulmonary valve disease (Cardiac disorders) | 1 (1) | 0 (0)
Restrictive cardiomyopathy (Cardiac disorders) | 0 (0) | 1 (1)
Right ventricular dysfunction (Cardiac disorders) | 1 (1) | 0 (0)
Sinus bradycardia (Cardiac disorders) | 1 (1) | 0 (0)
Sinus tachycardia (Cardiac disorders) | 3 (3) | 3 (3)
Supraventricular tachycardia (Cardiac disorders) | 0 (0) | 1 (1)
Tricuspid valve disease (Cardiac disorders) | 0 (0) | 1 (1)
Ventricular tachycardia (Cardiac disorders) | 1 (1) | 0 (0)
Congen, family, genetic disord -Oth spec (Congenital, familial and genetic disorders) | 1 (1) | 0 (0)
Ear and labyrinth disorders - Oth spec (Ear and labyrinth disorders) | 8 (8) | 4 (4)
Ear pain (Ear and labyrinth disorders) | 4 (4) | 2 (2)
External ear inflammation (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Hearing impaired (Ear and labyrinth disorders) | 0 (0) | 1 (1)
Middle ear inflammation (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Tinnitus (Ear and labyrinth disorders) | 3 (5) | 2 (2)
Vertigo (Ear and labyrinth disorders) | 13 (17) | 7 (8)
Vestibular disorder (Ear and labyrinth disorders) | 0 (0) | 2 (2)
Endocrine disorders - Other, specify (Endocrine disorders) | 0 (0) | 1 (1)
Hyperparathyroidism (Endocrine disorders) | 0 (0) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 2 (2) | 0 (0)
Hypothyroidism (Endocrine disorders) | 1 (1) | 0 (0)
Virilization (Endocrine disorders) | 1 (1) | 0 (0)
Blurred vision (Eye disorders) | 12 (22) | 4 (5)
Cataract (Eye disorders) | 2 (3) | 1 (1)
Dry eye (Eye disorders) | 13 (18) | 4 (4)
Eye disorders - Other, specify (Eye disorders) | 29 (41) | 9 (12)
Eye pain (Eye disorders) | 5 (5) | 1 (1)
Eyelid function disorder (Eye disorders) | 0 (0) | 1 (1)
Flashing lights (Eye disorders) | 2 (2) | 0 (0)
Floaters (Eye disorders) | 2 (2) | 0 (0)
Glaucoma (Eye disorders) | 1 (1) | 1 (1)
Keratitis (Eye disorders) | 1 (1) | 1 (1)
Periorbital edema (Eye disorders) | 1 (1) | 0 (0)
Photophobia (Eye disorders) | 1 (1) | 1 (1)
Uveitis (Eye disorders) | 1 (1) | 0 (0)
Watering eyes (Eye disorders) | 13 (16) | 5 (5)
Abdominal distension (Gastrointestinal disorders) | 1 (3) | 2 (2)
Abdominal pain (Gastrointestinal disorders) | 46 (58) | 16 (16)
Anal fistula (Gastrointestinal disorders) | 4 (4) | 0 (0)
Anal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Anal mucositis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Anal pain (Gastrointestinal disorders) | 5 (6) | 1 (3)
Anal ulcer (Gastrointestinal disorders) | 2 (2) | 0 (0)
Bloating (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cheilitis (Gastrointestinal disorders) | 2 (2) | 0 (0)
Colitis (Gastrointestinal disorders) | 3 (3) | 0 (0)
Constipation (Gastrointestinal disorders) | 33 (42) | 24 (32)
Dental caries (Gastrointestinal disorders) | 2 (3) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 182 (551) | 92 (166)
Dry mouth (Gastrointestinal disorders) | 7 (8) | 5 (5)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Dyspepsia (Gastrointestinal disorders) | 9 (10) | 6 (7)
Dysphagia (Gastrointestinal disorders) | 6 (6) | 2 (2)
Esophageal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophageal pain (Gastrointestinal disorders) | 0 (0) | 1 (1)
Esophageal ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Fecal incontinence (Gastrointestinal disorders) | 2 (2) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 1 (2)
Gastric ulcer (Gastrointestinal disorders) | 1 (1) | 0 (0)
Gastritis (Gastrointestinal disorders) | 11 (14) | 3 (7)
Gastroesophageal reflux disease (Gastrointestinal disorders) | 18 (22) | 9 (10)
Gastrointestinal disorders - Oth spec (Gastrointestinal disorders) | 33 (59) | 13 (19)
Gastrointestinal pain (Gastrointestinal disorders) | 6 (9) | 3 (6)
Gingival pain (Gastrointestinal disorders) | 1 (1) | 2 (2)
Hemorrhoidal hemorrhage (Gastrointestinal disorders) | 2 (3) | 1 (1)
Hemorrhoids (Gastrointestinal disorders) | 17 (19) | 6 (7)
Lip pain (Gastrointestinal disorders) | 2 (2) | 0 (0)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Mucositis oral (Gastrointestinal disorders) | 91 (235) | 17 (21)
Nausea (Gastrointestinal disorders) | 75 (132) | 40 (58)
Oral cavity fistula (Gastrointestinal disorders) | 1 (1) | 0 (0)
Oral pain (Gastrointestinal disorders) | 9 (15) | 6 (6)
Periodontal disease (Gastrointestinal disorders) | 2 (2) | 2 (2)
Rectal hemorrhage (Gastrointestinal disorders) | 9 (11) | 0 (0)
Rectal pain (Gastrointestinal disorders) | 2 (3) | 0 (0)
Stomach pain (Gastrointestinal disorders) | 6 (7) | 0 (0)
Tooth development disorder (Gastrointestinal disorders) | 2 (2) | 0 (0)
Toothache (Gastrointestinal disorders) | 3 (3) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 38 (68) | 21 (33)
Chills (General disorders) | 5 (5) | 2 (2)
Edema face (General disorders) | 3 (3) | 0 (0)
Edema limbs (General disorders) | 18 (23) | 15 (18)
Facial pain (General disorders) | 1 (1) | 0 (0)
Fatigue (General disorders) | 135 (346) | 96 (152)
Fever (General disorders) | 41 (60) | 14 (22)
Flu like symptoms (General disorders) | 21 (29) | 18 (35)
Gait disturbance (General disorders) | 2 (2) | 3 (3)
Gen disord and admin site conds-Oth spec (General disorders) | 44 (58) | 19 (27)
Injection site reaction (General disorders) | 5 (7) | 2 (3)
Localized edema (General disorders) | 8 (9) | 4 (6)
Malaise (General disorders) | 5 (7) | 3 (3)
Neck edema (General disorders) | 1 (1) | 1 (1)
Non-cardiac chest pain (General disorders) | 13 (14) | 7 (7)
Pain (General disorders) | 58 (120) | 62 (152)
Cholecystitis (Hepatobiliary disorders) | 2 (2) | 0 (0)
Hepatic pain (Hepatobiliary disorders) | 1 (1) | 1 (1)
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 6 (7) | 1 (1)
Portal vein thrombosis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Allergic reaction (Immune system disorders) | 4 (4) | 4 (4)
Autoimmune disorder (Immune system disorders) | 1 (1) | 0 (0)
Immune system disorders - Other, specify (Immune system disorders) | 3 (4) | 1 (1)
Bladder infection (Infections and infestations) | 1 (1) | 0 (0)
Bronchial infection (Infections and infestations) | 14 (17) | 7 (12)
Conjunctivitis (Infections and infestations) | 13 (16) | 5 (5)
Conjunctivitis infective (Infections and infestations) | 0 (0) | 1 (1)
Enterocolitis infectious (Infections and infestations) | 2 (2) | 0 (0)
Eye infection (Infections and infestations) | 2 (4) | 0 (0)
Gum infection (Infections and infestations) | 4 (4) | 1 (1)
Infections and infestations - Oth spec (Infections and infestations) | 83 (118) | 35 (51)
Laryngitis (Infections and infestations) | 3 (4) | 1 (1)
Lip infection (Infections and infestations) | 6 (7) | 0 (0)
Lung infection (Infections and infestations) | 11 (12) | 1 (1)
Mucosal infection (Infections and infestations) | 3 (3) | 0 (0)
Nail infection (Infections and infestations) | 15 (22) | 13 (14)
Otitis externa (Infections and infestations) | 1 (1) | 2 (2)
Otitis media (Infections and infestations) | 1 (1) | 1 (1)
Papulopustular rash (Infections and infestations) | 6 (7) | 2 (2)
Paronychia (Infections and infestations) | 9 (9) | 7 (9)
Peripheral nerve infection (Infections and infestations) | 1 (1) | 0 (0)
Pharyngitis (Infections and infestations) | 5 (5) | 2 (2)
Phlebitis infective (Infections and infestations) | 1 (1) | 0 (0)
Rash pustular (Infections and infestations) | 5 (5) | 1 (1)
Rhinitis infective (Infections and infestations) | 4 (4) | 1 (1)
Salivary gland infection (Infections and infestations) | 1 (1) | 0 (0)
Sinusitis (Infections and infestations) | 15 (17) | 5 (7)
Skin infection (Infections and infestations) | 26 (46) | 14 (22)
Small intestine infection (Infections and infestations) | 0 (0) | 1 (1)
Soft tissue infection (Infections and infestations) | 1 (1) | 1 (1)
Tooth infection (Infections and infestations) | 10 (11) | 4 (4)
Tracheitis (Infections and infestations) | 2 (2) | 1 (1)
Upper respiratory infection (Infections and infestations) | 38 (52) | 24 (36)
Urinary tract infection (Infections and infestations) | 26 (57) | 20 (32)
Uterine infection (Infections and infestations) | 1 (2) | 0 (0)
Vaginal infection (Infections and infestations) | 8 (12) | 2 (2)
Ankle fracture (Injury, poisoning and procedural complications) | 3 (3) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 10 (12) | 2 (3)
Dermatitis radiation (Injury, poisoning and procedural complications) | 0 (0) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 15 (26) | 9 (15)
Fracture (Injury, poisoning and procedural complications) | 14 (16) | 4 (5)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Infusion related reaction (Injury, poisoning and procedural complications) | 2 (2) | 1 (1)
Inj, pois and proced complic - Oth spec (Injury, poisoning and procedural complications) | 2 (2) | 3 (5)
Radiation recall reaction (dermatologic) (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Seroma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Spinal fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1) | 1 (1)
Wound complication (Injury, poisoning and procedural complications) | 1 (2) | 2 (2)
Wrist fracture (Injury, poisoning and procedural complications) | 3 (3) | 2 (2)
Activated partial throm time prolonged (Investigations) | 2 (2) | 0 (0)
Alanine aminotransferase increased (Investigations) | 32 (63) | 9 (11)
Alkaline phosphatase increased (Investigations) | 13 (21) | 7 (9)
Aspartate aminotransferase increased (Investigations) | 33 (63) | 10 (12)
Blood bilirubin increased (Investigations) | 5 (6) | 3 (5)
Cholesterol high (Investigations) | 5 (5) | 6 (6)
Creatinine increased (Investigations) | 14 (29) | 8 (10)
Ejection fraction decreased (Investigations) | 22 (32) | 28 (51)
Forced expiratory volume decreased (Investigations) | 1 (1) | 1 (2)
GGT increased (Investigations) | 3 (5) | 2 (3)
Investigations - Other, specify (Investigations) | 15 (60) | 6 (16)
Lipase increased (Investigations) | 0 (0) | 1 (2)
Lymphocyte count decreased (Investigations) | 32 (145) | 10 (37)
Neutrophil count decreased (Investigations) | 196 (1618) | 20 (32)
Platelet count decreased (Investigations) | 59 (174) | 4 (7)
Weight gain (Investigations) | 6 (12) | 6 (7)
Weight loss (Investigations) | 11 (14) | 6 (21)
White blood cell decreased (Investigations) | 98 (613) | 10 (31)
Anorexia (Metabolism and nutrition disorders) | 34 (50) | 12 (14)
Dehydration (Metabolism and nutrition disorders) | 6 (7) | 4 (4)
Hypercalcemia (Metabolism and nutrition disorders) | 3 (3) | 4 (6)
Hyperglycemia (Metabolism and nutrition disorders) | 16 (30) | 10 (31)
Hyperkalemia (Metabolism and nutrition disorders) | 3 (4) | 3 (3)
Hypernatremia (Metabolism and nutrition disorders) | 5 (6) | 0 (0)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (2) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 10 (12) | 2 (6)
Hypocalcemia (Metabolism and nutrition disorders) | 19 (30) | 7 (18)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (3) | 2 (2)
Hypokalemia (Metabolism and nutrition disorders) | 40 (78) | 13 (21)
Hypomagnesemia (Metabolism and nutrition disorders) | 12 (25) | 4 (4)
Hyponatremia (Metabolism and nutrition disorders) | 6 (8) | 3 (3)
Hypophosphatemia (Metabolism and nutrition disorders) | 3 (3) | 1 (2)
Metabolism, nutrition disord - Oth spec (Metabolism and nutrition disorders) | 4 (4) | 4 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 66 (97) | 85 (145)
Arthritis (Musculoskeletal and connective tissue disorders) | 11 (16) | 6 (7)
Back pain (Musculoskeletal and connective tissue disorders) | 27 (38) | 29 (33)
Bone pain (Musculoskeletal and connective tissue disorders) | 21 (26) | 15 (17)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3)
Flank pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 1 (1)
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 13 (14) | 5 (6)
Joint effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2)
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (5)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 5 (12) | 2 (2)
Muscle weakness trunk (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1)
Muscle weakness upper limb (Musculoskeletal and connective tissue disorders) | 2 (2) | 1 (1)
Musculoskeletal deformity (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Musculoskeletal, conn tissue - Oth spec (Musculoskeletal and connective tissue disorders) | 51 (69) | 38 (58)
Myalgia (Musculoskeletal and connective tissue disorders) | 27 (37) | 29 (37)
Neck pain (Musculoskeletal and connective tissue disorders) | 7 (7) | 5 (5)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 4 (4) | 4 (4)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 4 (4) | 6 (6)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 33 (55) | 21 (30)
Neoplasms benign, mal, uncpec - Oth spec (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (6) | 3 (4)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Amnesia (Nervous system disorders) | 1 (1) | 1 (1)
Aphonia (Nervous system disorders) | 1 (1) | 0 (0)
Central nervous system necrosis (Nervous system disorders) | 1 (1) | 0 (0)
Cognitive disturbance (Nervous system disorders) | 3 (3) | 4 (4)
Concentration impairment (Nervous system disorders) | 4 (4) | 1 (2)
Depressed level of consciousness (Nervous system disorders) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 37 (50) | 21 (27)
Dysarthria (Nervous system disorders) | 0 (0) | 1 (1)
Dysesthesia (Nervous system disorders) | 3 (3) | 3 (3)
Dysgeusia (Nervous system disorders) | 10 (12) | 5 (6)
Dysphasia (Nervous system disorders) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 65 (86) | 46 (67)
Hypersomnia (Nervous system disorders) | 2 (2) | 0 (0)
Lethargy (Nervous system disorders) | 2 (2) | 0 (0)
Memory impairment (Nervous system disorders) | 4 (5) | 6 (6)
Movements involuntary (Nervous system disorders) | 1 (1) | 1 (1)
Muscle weakness left-sided (Nervous system disorders) | 1 (5) | 0 (0)
Muscle weakness right-sided (Nervous system disorders) | 1 (1) | 0 (0)
Nervous system disorders - Oth spec (Nervous system disorders) | 11 (11) | 13 (17)
Neuralgia (Nervous system disorders) | 3 (3) | 2 (2)
Olfactory nerve disorder (Nervous system disorders) | 1 (1) | 0 (0)
Paresthesia (Nervous system disorders) | 19 (21) | 8 (10)
Peripheral motor neuropathy (Nervous system disorders) | 10 (10) | 11 (14)
Peripheral sensory neuropathy (Nervous system disorders) | 50 (59) | 28 (38)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1)
Seizure (Nervous system disorders) | 3 (4) | 1 (1)
Somnolence (Nervous system disorders) | 2 (2) | 1 (1)
Spasticity (Nervous system disorders) | 0 (0) | 1 (1)
Stroke (Nervous system disorders) | 0 (0) | 1 (1)
Syncope (Nervous system disorders) | 3 (6) | 3 (3)
Tremor (Nervous system disorders) | 3 (3) | 1 (1)
Agitation (Psychiatric disorders) | 0 (0) | 3 (3)
Anxiety (Psychiatric disorders) | 14 (18) | 17 (19)
Confusion (Psychiatric disorders) | 3 (6) | 0 (0)
Depression (Psychiatric disorders) | 7 (7) | 8 (9)
Hallucinations (Psychiatric disorders) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 30 (42) | 29 (31)
Irritability (Psychiatric disorders) | 1 (2) | 2 (2)
Libido decreased (Psychiatric disorders) | 2 (2) | 1 (1)
Personality change (Psychiatric disorders) | 1 (1) | 0 (0)
Psychiatric disorders - Other, specify (Psychiatric disorders) | 7 (9) | 9 (10)
Restlessness (Psychiatric disorders) | 0 (0) | 1 (1)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Bladder spasm (Renal and urinary disorders) | 0 (0) | 1 (1)
Cystitis noninfective (Renal and urinary disorders) | 4 (5) | 1 (1)
Hematuria (Renal and urinary disorders) | 4 (4) | 2 (2)
Hemoglobinuria (Renal and urinary disorders) | 0 (0) | 1 (1)
Renal and urinary disorders - Oth spec (Renal and urinary disorders) | 6 (7) | 4 (4)
Renal calculi (Renal and urinary disorders) | 2 (3) | 0 (0)
Renal colic (Renal and urinary disorders) | 0 (0) | 2 (2)
Urinary frequency (Renal and urinary disorders) | 4 (4) | 4 (4)
Urinary incontinence (Renal and urinary disorders) | 5 (6) | 3 (4)
Urinary retention (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary tract pain (Renal and urinary disorders) | 6 (7) | 2 (2)
Urinary urgency (Renal and urinary disorders) | 3 (4) | 1 (1)
Breast pain (Reproductive system and breast disorders) | 10 (12) | 7 (7)
Dysmenorrhea (Reproductive system and breast disorders) | 0 (0) | 1 (2)
Dyspareunia (Reproductive system and breast disorders) | 8 (8) | 3 (3)
Menorrhagia (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Pelvic pain (Reproductive system and breast disorders) | 2 (2) | 2 (3)
Reproductive system and breast -Oth spec (Reproductive system and breast disorders) | 7 (7) | 3 (3)
Uterine hemorrhage (Reproductive system and breast disorders) | 0 (0) | 1 (1)
Uterine pain (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal discharge (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Vaginal dryness (Reproductive system and breast disorders) | 28 (31) | 10 (11)
Vaginal hemorrhage (Reproductive system and breast disorders) | 4 (4) | 4 (4)
Vaginal inflammation (Reproductive system and breast disorders) | 3 (3) | 1 (1)
Vaginal pain (Reproductive system and breast disorders) | 1 (2) | 1 (1)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 18 (20) | 9 (9)
Aspiration (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchial obstruction (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 39 (55) | 28 (36)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 26 (37) | 25 (36)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 46 (59) | 13 (14)
Hoarseness (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Laryngeal hemorrhage (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (2)
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 0 (0)
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 19 (20) | 7 (7)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (2)
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 5 (6) | 0 (0)
Productive cough (Respiratory, thoracic and mediastinal disorders) | 6 (7) | 4 (6)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Resp, thoracic, mediastinal - Oth spec (Respiratory, thoracic and mediastinal disorders) | 24 (36) | 8 (11)
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Sinus pain (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Sleep apnea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Sneezing (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Sore throat (Respiratory, thoracic and mediastinal disorders) | 16 (26) | 7 (7)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Wheezing (Respiratory, thoracic and mediastinal disorders) | 2 (3) | 0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 28 (30) | 9 (10)
Bullous dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Dry skin (Skin and subcutaneous tissue disorders) | 23 (30) | 13 (18)
Erythema multiforme (Skin and subcutaneous tissue disorders) | 6 (6) | 7 (8)
Erythroderma (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (2)
Hirsutism (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Nail discoloration (Skin and subcutaneous tissue disorders) | 9 (10) | 5 (5)
Nail loss (Skin and subcutaneous tissue disorders) | 9 (9) | 5 (6)
Nail ridging (Skin and subcutaneous tissue disorders) | 9 (9) | 8 (8)
Pain of skin (Skin and subcutaneous tissue disorders) | 1 (1) | 2 (2)
Palmar-plantar erythrodysesthesia syndrm (Skin and subcutaneous tissue disorders) | 3 (4) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 55 (95) | 42 (60)
Purpura (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2)
Rash acneiform (Skin and subcutaneous tissue disorders) | 19 (24) | 12 (16)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 24 (39) | 26 (29)
Scalp pain (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (2)
Skin and subcut tissue disord - Oth spec (Skin and subcutaneous tissue disorders) | 63 (128) | 36 (65)
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Skin hypopigmentation (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
Skin ulceration (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1)
Urticaria (Skin and subcutaneous tissue disorders) | 3 (3) | 2 (4)
Surgical and medical proced - Oth spec (Surgical and medical procedures) | 3 (3) | 3 (4)
Capillary leak syndrome (Vascular disorders) | 0 (0) | 1 (1)
Flushing (Vascular disorders) | 3 (3) | 8 (9)
Hematoma (Vascular disorders) | 4 (4) | 3 (3)
Hot flashes (Vascular disorders) | 55 (91) | 63 (81)
Hypertension (Vascular disorders) | 21 (37) | 21 (28)
Hypotension (Vascular disorders) | 4 (5) | 2 (3)
Lymphedema (Vascular disorders) | 10 (13) | 6 (6)
Lymphocele (Vascular disorders) | 1 (1) | 0 (0)
Phlebitis (Vascular disorders) | 1 (1) | 0 (0)
Superficial thrombophlebitis (Vascular disorders) | 1 (1) | 1 (1)
Thromboembolic event (Vascular disorders) | 6 (7) | 8 (10)
Vascular disorders - Other, specify (Vascular disorders) | 8 (17) | 5 (10)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-02-09): https://cdn.clinicaltrials.gov/large-docs/85/NCT02947685/Prot_SAP_000.pdf